CLINICAL TRIAL: NCT01547169
Title: Study of Nasal Insulin to Fight Forgetfulness - Long-acting Insulin Detemir - 21 Days
Acronym: SNIFF-LONG 21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Suzanne Craft, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39683-A; 2P50AG005136-27 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-03-07 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: memory; intranasal insulin; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator)
  Interventions: Drug: Placebo Comparator
- Low Dose Insulin Detemir (10IU bid) (Experimental)
  Interventions: Drug: insulin detemir
- High Dose Insulin Detemir (20IU bid) (Experimental)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: Placebo Comparator — saline, taken twice per day for a 3 week duration
  Arms: Saline
Drug: insulin detemir — 10IU of insulin detemir, administered intranasally twice per day for a 3 week duration
  Other Names: Levemir
  Arms: Low Dose Insulin Detemir (10IU bid)
Drug: insulin detemir — 20IU insulin detemir, administered intranasally twice per day for a 3 week duration
  Other Names: Levemir
  Arms: High Dose Insulin Detemir (20IU bid)

SUMMARY:
The study will examine the effects of intranasally administered long-acting insulin detemir on cognition in persons with Alzheimer's disease (AD) or amnestic mild cognitive impairment (aMCI). The rationale for these studies is derived from growing evidence that insulin contributes to multiple brain functions, and that insulin dysregulation can contribute to AD pathogenesis. Thus, therapies aimed at restoring normal insulin signaling in the CNS may have beneficial effects on brain function. Intranasal administration of insulin increases insulin signaling in brain without raising peripheral levels and causing hypoglycemia. Insulin detemir is an insulin analogue that may have better action in brain than other insulin formulations because of its albumin binding properties. The investigators will test the therapeutic effects of intranasally-administered insulin detemir in a dose-finding study in which participants will receive one of two doses of insulin detemir or placebo for a three week period. The investigators will test the hypothesis that either dose will improve memory and daily functioning in persons with AD/aMCI compared with placebo.

DETAILED DESCRIPTION:
It is well-known that insulin, a hormone that is naturally secreted by the pancreas, plays an important physiological role by regulating blood sugar levels in the body. The investigators now know that insulin plays many important roles in the brain as well. Insulin seems to be especially active in the part of the brain that corresponds to learning and memory. Studies have shown that when people have insufficient insulin in the brain (which, for example, is the case with Type-II diabetes), they are increasingly at risk to develop memory problems and Alzheimer's disease. In a past study, the investigators administered intravenous insulin to participants and found that it improves their memory. However, that particular method would not be a practical intervention for people with Alzheimer's disease due to the risk of hypoglycemia or exacerbation of insulin resistance. Instead, the investigators use an "intranasal" method of administration, in which the insulin is inserted into a device, and administered intranasally. In this method, the insulin travels directly to the brain, and bypasses the body. Our past studies have also demonstrated that this can be a reliable way to improve memory, and it does not change the body's blood glucose levels.

In our past studies, the investigators have used regular insulin, which lasts about 3-4 hours and creates a similar "spike" in insulin that one would have after eating a meal. However, in normal physiology, the pancreas also releases small and more constant "pulses" of insulin throughout the day and night, establishing a base level of insulin. Accordingly, several longer-lasting types of insulin are now available that last closer to 10-12 hours, mimicking that base level of insulin. The current study uses a long-lasting type of insulin called "insulin detemir," to determine if learning and memory will benefit from a more constant supplement of insulin. the investigators want to determine whether this treatment can benefit people who already have a memory impairment-either they already have a diagnosis of Alzheimer's disease or are diagnosed with mild cognitive impairment, a condition that precedes Alzheimer's disease, and whether a lower or higher dose of insulin detemir is more effective. The investigators will examine cognition, daily function, and different markers of Alzheimer's disease that are in the blood as outcome measures.

The investigators have these specific aims:

1. The investigators will test the hypothesis that compared to placebo, three weeks of treatment with intranasal insulin detemir will improve cognition and function in adults with Alzheimer's Disease (AD) or Mild Cognitive Impairment (MCI).
2. The investigators will determine which of two doses of intranasal insulin detemir produces the greatest improvement in cognition and daily function relative to placebo for adults with AD or MCI.

To examine these hypotheses, the investigators are recruiting approximately 60 participants who have been diagnosed with AD or MCI. They will be randomly selected to take a lower dose of insulin detemir, a higher dose of insulin detemir, or saline (which is an inactive substance and will serve as a placebo). Cognition and the level of daily function will be tested before they begin the study drug, and after 3 weeks of the study drug. The investigators will also measure glucose tolerance and take blood samples to measure markers of AD in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-89
* Diagnosed with mild cognitive impairment, or mild/moderate AD

Exclusion Criteria:

* Excessively high or low blood pressure, heart rate
* BMI greater than 34
* Pre-existing diabetes not controlled by exercise
* Previous/current use of insulin
* Significant elevations in lipids, liver enzymes
* Menstrual period within the last 12 months
* Significant neurological or medical disorder (other than AD)
* Significant use of nasal decongestants
* Current use of anti-psychotic, anti-convulsive, anxiolytic, glucocorticoids, or sedative medications

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Verbal Memory Composite | Change from Baseline in Verbal Memory at 3 Weeks
  The composite will consist of the weighted sum of Immediate + Delayed Story Recall and Immediate +Delayed List Recall

SECONDARY OUTCOMES:
Neuropsychological Test of Executive Function 1 | Change from Baseline in Executive Functioning at 3 Weeks
  Computerized Dot Counting Test (test of executive functioning)
Glucose Tolerance | Change from Baseline in Glucose Tolerance at 3 Weeks
  Subjects will undergo oral glucose tolerance test (OGTT) to assess glucose tolerance
Functional Ability | Change from Baseline in Functional Ability at 3 Weeks
  Subjects will have a collateral informant (i.e., spouse or friend) rate the subjects' ability to carry out activities of daily living on the Dementia Severity Rating Scale.
Plasma biomarkers of AD | Change from Baseline in Plasma Biomarkers at 3 Weeks
  Plasma Abeta (ABeta 38, ABeta 40, and Abeta 42) and Tau (total tau and phosphorylated tau) will be measured in each subject.
Neuropsychological Test of Executive Functioning 2 | Change from Baseline in Executive Functioning at 3 Weeks
  Computerized Stroop Test
Neuropsychological Tests of Visual Working Memory | Change from Baseline in Visual Working Memory at 3 Weeks
  Benton Visual Retention Test Form F&G (a test of visual working memory)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — VA Puget Sound Health Care System; University of Washington School of Medicine
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States